CLINICAL TRIAL: NCT02673229
Title: Comparison of Collagenase Santyl Ointment With Antibiotic Ointment in the Outpatient Care of Minor Partial Thickness Burns
Brief Title: Comparison of Collagenase With Antibiotic Ointment of Minor Partial Thickness Burns
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: slow enrollment due to cost of medication and conflict of interest enrolling uninsured patients
Sponsor: University of Kansas Medical Center (Other)
Responsible Party: Principal Investigator, Dhaval Bhavsar, Assistant Professor, University of Kansas Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13663
Record Dates: First submitted 2016-02-01; First posted 2016-02-03 (Estimated); Results first posted 2024-07-10 (Actual); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Burn, Partial Thickness
Keywords: Santyl; Burn; Partial Thickness Burn; Second Degree Burn; Minor Burn Bacitracin; Scar Appearance
MeSH Terms: conditions — Burns | interventions — Bacitracin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Collagenase Santyl (Active Comparator): Applied topically (2 mm thickness once daily)
  Interventions: Drug: Collagenase Santyl
- Bacitracin (Sham Comparator): Applied topically (2 mm thickness) once daily
  Interventions: Drug: Bacitracin

INTERVENTIONS:
Drug: Collagenase Santyl — A sterile, enzymatic debriding agent which contains 250 collagenase units per gram of white petrolatum, United States Pharmacopeia (USP).
  Arms: Collagenase Santyl
Drug: Bacitracin — One gram is equal to 500 bacitracin units; one unit of bacitracin is equivalent to 0.026 milligrams.
  Other Names: Bacitracin Zinc Ointment
  Arms: Bacitracin

SUMMARY:
By doing this study, researchers hope to learn if applying Santyl to the burn during the healing process affects the appearance of the resulting scar.

DETAILED DESCRIPTION:
Subjects who have minor, second degree burns may be enrolled in this study. Subjects will receive either Santyl ointment or bacitracin ointment to apply to the burn until it heals. Bandages will be used to keep the burn covered while it heals. Second degree burns generally leave a scar. Once the burn heals, lotion and an appropriate bandage will be used to try to minimize the appearance of a scar.

The study hypothesis is that burns treated with Santyl will have a better scar appearance than burns treated with bacitracin.

Subjects enrolled in this study will make once a week visits to the University of Kansas Medical Center outpatient burn clinic until the burn heals. The burn will be assessed for healing at these visits. Once healed, visits to the clinic will be at 60 & 180 days, up to 6 months. At these visits, the appearance of the scar will be evaluated.

This study was originally funded by Smith and Nephew, but Smith and Nephew is no longer providing support for the study.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent, which will consist of reading, signing, and dating the informed consent document after the Investigator, sub-Investigator or other designated study staff member has explained the study procedures, risks, and contact information. For subjects not able to provide informed consent (e.g., minors), a parent or legally authorized representative must provide consent. Assent must be provided as required by the Institutional Review Board (IRB).
2. Have one or more acute burns which:

   1. are thermal, chemical or electrical in etiology
   2. in aggregate cover <10% total body surface area (TBSA)
   3. are each equal to or less than 72 hrs old
   4. are each no more than deep partial thickness (2nd degree)
   5. are not visibly infected
3. Able to take in oral fluids.
4. Able to comply with the requirement for daily dressing changes, or have a caretaker who is able to comply.
5. Willing to make all required study visits.

Exclusion Criteria:

1. Contraindications or hypersensitivity to the use of the test article or their components (e.g., known hypersensitivity to bacitracin).
2. Embedded foreign bodies in the burn wound which cannot be immediately removed.
3. The burned tissue includes or is within 1 cm of the eye or genitalia.
4. Severe perioral burns.
5. Airway involvement or aspiration of hot liquids.
6. Suspicion of physical abuse.
7. Burn wound requires a skin graft.
8. Outpatient management of the burn wound is not appropriate.
9. Participation in another investigational clinical study within thirty (30) days of the Screening Visit.
10. The Investigator may declare any subject ineligible for a valid medical reason. Current or recent (< 6 months) history of severe, unstable, or uncontrolled neurological, cardiovascular, gastrointestinal, hematological, hepatic, and/or renal disease or evidence of other diseases based upon a review of medical history that, in the opinion of the Investigator, would preclude safe subject participation in the study.
11. Test articles are cost-prohibitive for subjects

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2018-12-27 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dhaval Bhavsar, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- See also: Initial study registration by study agent manufacturer before the study was modified and taken over by a new sponsor — http://clinicaltrials.gov/ct2/show/NCT01516463

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Collagenase Santyl | Bacitracin
Started | 8 | 12
Completed | 7 | 9
Not Completed | 1 | 3

BASELINE CHARACTERISTICS:
Population: This is descriptive statistics on the demographic information for each group, the bacitracin group and the santyl group.
Groups:
- Total: Total of all reporting groups
Arm/Group | Collagenase Santyl | Bacitracin | Total
Number analyzed (Participants) | 8 | 12 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 7 | 12 | 19
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 38 [12 to 56] | 36 [19 to 48] | 37 [12 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 5
  Male | 6 | 9 | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 6 | 10 | 16
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 12 | 20
Fitzpatrick Skin Type [Count of Participants; unit: Participants] — The Fitzpatrick skin classification is a measure of a person's skin pigment and propensity to form a hypertrophic scar. Lower Fitzpatrick Skin scores indicate a person's propensity to burn easily or scar easily.
  Type 1: Light, pale white, always burns, never tans. Type 2: Fair, white. Usually burns, sometimes tans. Type 3: Medium to olive. Sometimes burns, usually tans. Type 4: Olive. Rarely burns, always tans. Type 5: Brown, very rarely burns, always tans. Type 6: Dark brown to black, Never burns, always tans.
  Participants
    Type 2 | 1 | 2 | 3
    Type 3 | 3 | 6 | 9
    Type 4 | 2 | 3 | 5
    Type 5 | 0 | 0 | 0
    Type 6 | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With at Least 95% Wound Healing
Description: Outcome will be reported as number of subjects with at least 95% wound healing
Time Frame: 21 Days After Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Santyl | Bacitracin
Number analyzed (Participants) | 8 | 12
Participants | 6 | 7

2. Primary Outcome: Number of Subjects With at Least 95% Wound Healing
Description: Outcome will be reported as number of subjects with at least 95% wound epithelialization
Time Frame: 14 days after treatment
Population: number of participants healed after 14 days of treatment
Measure: Count of Participants; unit: Participants
Groups:
- Collagenase; Bacitracin: Apply topically 2mm thick
Arm/Group | Collagenase | Bacitracin
Number analyzed (Participants) | 8 | 12
Participants | 4 | 5

3. Secondary Outcome: Vancouver Scar Scale
Description: Scar appearance will be documented using the Vancouver Scar Scale. It assesses 4 variables: vascularity, height/thickness, pliability, and pigmentation. VSS is derived by adding the score for each variable. Details of VSS is below.
  The Vancouver Scar Scale
  Pigmentation (0-2) Normal 0 Hypopigmentation 1 Hyperpigmentation 2 Range of Score: 0-2 with 0 = best outcome, 2 = worst outcome
  Vascularity (0-3) Normal. 0 Pink 1 Red 2 Purple. 3 Range: 0-3 with 0 = best outcome, 3 = worst outcome
  Pliability (0-5) Normal 0 Supple 1 Yielding 2 Firm 3 Banding 4 Contracture 5 Range of Score: 0-5, with 0 = best outcome, 5 = worst outcome
  Height (0-3) Normal (flat) 0 0-2 mm 1 2-5 mm 2 >5 mm 3 Range of Score 0-3, with 0 = best outcome, 3 = worst outcome
  Interpretation of Total Score: 0 = best outcome, 13 = worst outcome
Time Frame: 90 Days After Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Santyl | Bacitracin
Number analyzed (Participants) | 6 | 2
Participants
  Score of 0 | 2 | 1
  Score of 2 | 1 | 1
  Score of 4 | 2 | 0
  Score of 8 | 1 | 0

4. Other Pre Specified Outcome: Time to Healing
Description: time to heal in days
Time Frame: Up To 90 Days After Treatment
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Collagenase Santyl | Bacitracin
Number analyzed (Participants) | 8 | 12
days | 18.67 (6.6) | 28.22 (24.5)

5. Other Pre Specified Outcome: Number of Participants With a Burn Wound Infection
Description: Number of participants with a burn wound infection cellulitis
Time Frame: Up to 90 Days After Treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Collagenase Santyl | Bacitracin
Number analyzed (Participants) | 8 | 12
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: During course of the study, over 90 days
Arm/Group | Collagenase Santyl | Bacitracin
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/12
Other Adverse Events (participants affected / at risk) | 1/8 | 3/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Collagenase Santyl (N=8) | Bacitracin (N=12)
rash (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) — dermatitis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-07): https://cdn.clinicaltrials.gov/large-docs/29/NCT02673229/Prot_SAP_000.pdf